CLINICAL TRIAL: NCT03113591
Title: Evaluate the Effect of Osteo Introducer System in Total Hip Arthroplasty: A Prospective, Multicenter, Randomized Controlled Study
Brief Title: Evaluate the Effect of Osteo Introducer System in Total Hip Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Suzhou MicroPort OrthoRecon Co. LTD (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MP-GJ15-01
Record Dates: First submitted 2017-04-04; First posted 2017-04-13 (Actual); Last update posted 2019-04-04 (Actual); Status verified 2019-04

CONDITIONS: Joint Disease
Keywords: total hip arthroplasty; minimal invasive
MeSH Terms: conditions — Joint Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Osteo introducer group (Experimental): undergo minimal invasive total hip arthroplasty surgery
  Interventions: Procedure: Minimum invasive total hip arthroplasty
- Control group (Active Comparator): undergo common total hip arthroplasty surgery
  Interventions: Procedure: Common total hip arthroplasty

INTERVENTIONS:
Procedure: Minimum invasive total hip arthroplasty — Minimum invasive total hip arthroplasty using the osteo introducer system
  Arms: Osteo introducer group
Procedure: Common total hip arthroplasty — Common total hip arthroplasty using common instruments
  Arms: Control group

SUMMARY:
Osteo introducer system is the instruments used in minimal invasive THA. This study will compare the minimal invasive THA using the osteo introducer system and THA using common instruments, to show the non-inferiority of osteo introducer system in safety and efficacy of THA surgery.

ELIGIBILITY:
Inclusion Criteria:

* With indications of total hip arthroplasty (e.g. non-inflammatory degenerative joint disease such as osteoarthritis, avascular necrosis, ankylosis; rheumatoid arthritis; correction of functional deformity, etc.)
* BMI<30
* Subject is a candidate for primary total hip arthroplasty
* No obvious congenital abnormality in hip joint
* Subject has no mental illness, is willing to join the study voluntarily and sign the approved informed consent document; is willing and able to complete required study visits or assessments

Exclusion Criteria:

* Subjects with inadequate neuromuscular status (e.g., prior paralysis, fusion and/or inadequate abductor strength), poor bone stock, poor skin coverage around the joint which would make the procedure unjustifiable
* Overt infection
* Distant foci of infections
* Allergy to metals
* Rapid disease progression as manifested by joint destruction or bone absorption apparent on X-ray
* Skeletally immature
* Neuropathic joints
* Hepatitis or HIV infection
* Neurological or musculoskeletal disease that may adversely affect gait or weight-bearing
* Pregnant or lactating women
* Subjects enrolled in another drug or device clinical investigation within 3 month
* Investigator has judged the subject is not suitable for the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-08-29 (Actual); Primary Completion 2018-09-13 (Actual); Study Completion 2019-01-03 (Actual)

PRIMARY OUTCOMES:
Evaluation the restoration of hip function at 3 month | 3 month
  Assessment the changes of Harris Hip Score at postoperative 3 month from preoperative

SECONDARY OUTCOMES:
Evaluation of X-ray | 1day, 6 week, 6 month
  Assessment of position, confirm whether there is loosening, dislocation or fracture etc.
Evaluation the restoration of hip function at each time frame | 6 week, 3 month, 6 month
  Assessment the Harris Hip Score at each time frame
Barthel Index | 1day, 3day, 2 week, 6 week, 3 month, 6 month
  Assessment the daily living activity
Berg Balance Scale | 1day, 3day, 2 week, 6 week, 3 month, 6 month
  Assessment the balance ability
Visual Analogue Scale | 1day, 3day, 2 week
  Assessment the degree of pain
The use of analgesics | 1day, 3day, 2 week, 6 week, 3 month, 6 month
  Investigate the name and dosage of analgesics to indirectly assess the degree of pain
Adverse events | up to 6 month
  Investigate all the adverse events happened during the study period
Laboratory Examinations | 3 day, 6 week
  Collect the following laboratory results which reflect the traumatic stress:Glu, CRP, Alb, CK, TBA, UA, Ca, Mg, WBC, GRA
Dislocation rate | 1day, 3day, 2 week, 6 week, 3 month, 6 month
  Compare the dislocation rate

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Sixth People's Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No